CLINICAL TRIAL: NCT02854384
Title: Mobile Phone Radiation and Brain Rhythm in Epileptic Patients
Status: Completed | Type: Observational
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Noha El Sawy, Assistant Lecturer, Kasr El Aini Hospital
Other Study IDs: 1
Record Dates: First submitted 2016-07-31; First posted 2016-08-03 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Epilepsy
Keywords: Epilepsy; Mobile phone
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Epilepsy Patients: males and females whose age more than 18 years, diagnosed with epilepsy, regardless of whether symptomatic,idiopathic ,focal or generalized
- Healthy Control: males and females whose age more than 18 years

SUMMARY:
This work is intended to assess the effect of -30 minutes- exposure to mobile-phone on the functions of the central nervous system (CNS) in epileptic patients.

DETAILED DESCRIPTION:
This work shows the effect of the 30 minutes mobile waves' radiation over the normal person brain activity (EEG) and cognition (P300) together with the effect over the unstable brain of the epileptic patients. Exposure to mobile-phone radiation has been reported to increase the spectral power of electroencephalograms (EEGs), particularly in the alpha band, during both the waking and sleeping states. The tendency toward electrical instability of the neural networks of epileptic patients suggests that these individuals may be especially sensitive to electromagnetic fields espcially mobile-phone radiation (MPR). The short-term effects of exposure to electromagnetic (EM) fields on a number of cognitive variables such as memory, attention and speed of decision-making could be assedsed by P 300 latency and amplitude.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Above 18 years
* Epileptic patients (regardless of whether symptomatic, idiopathic, focal or generalized)

Exclusion Criteria:

* Age less than 18 years
* Chronic medical condition
* Epileptic fit in the last 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study included 30 epileptic patients and 30 healthy volunteers, males and females whose age above 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Digital Electroencephalography (EEG) examination | one day
P300 test | one day
  The P300 Test: Neurophysiological Test. P300 wave was defined as the most positive point of the average waveform to the target tones after 250 msec and before 600 msec. For each subject P300 latency and P300 amplitude were obtained to detect any significant abnormality

IPD SHARING:
Plan to Share IPD: Undecided